CLINICAL TRIAL: NCT01626638
Title: Clinical Evaluation of Confocal Microscopy in Head and Neck Cancer
Brief Title: Confocal Micro-endoscopy in Head and Neck Cancer/Micro Endoscopie Confocale (MEC)Oto-Rhino-Laryngologie (ORL)
Acronym: MEC ORL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00818-33
Record Dates: First submitted 2012-06-15; First posted 2012-06-25 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Malignant Pharyngo Laryngeal Tumors; Pre-malignant Pharyngo Laryngeal Tumors
Keywords: Patients with malignant and pre-malignant pharyngo laryngeal tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Procedure: Confocal Micro Endoscopy

INTERVENTIONS:
Procedure: Confocal Micro Endoscopy

SUMMARY:
The primary objective is to validate the diagnostic correlation between the intraoperative microendoscopic images and the conventional histological analysis on biopsy and/or surgical specimens on patients with epidermoid carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant and pre-malignant pharyngo laryngeal tumors in whom direct laryngoscopy was performed under general anesthesia with biopsies for diagnostic or endoscopic removal
* > 18 years
* signed ICF

Exclusion Criteria:

* Persons deprived of liberty
* Patients with history of allergy to patent blue
* Pregnant women or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Diagnostic correlation between confocal micro endoscopy and conventional histology | at an average of 18 months

SECONDARY OUTCOMES:
Histological diagnostic with confocal micro endoscopy (MEC) VS conventional histological analysis | At the time of the biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane TEMAM, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (2):
- France (2):
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Institut Universitaire Du Cancer de Toulouse - Oncopole, Toulouse

REFERENCES:
- [Derived] Villard A, Breuskin I, Casiraghi O, Asmandar S, Laplace-Builhe C, Abbaci M, Moya Plana A. Confocal laser endomicroscopy and confocal microscopy for head and neck cancer imaging: Recent updates and future perspectives. Oral Oncol. 2022 Apr;127:105826. doi: 10.1016/j.oraloncology.2022.105826. Epub 2022 Mar 19. PMID 35316771